CLINICAL TRIAL: NCT02533986
Title: Effects of Berry Peel Intake on Glucose Metabolism in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Elin Östman, Assoc. Prof., PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: COGBERRY-BR
Record Dates: First submitted 2015-08-20; First posted 2015-08-27 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Berry; Inflammation; Cognition; Polyphenols; Appetite; Glucose metabolism
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control drink (Placebo Comparator): Dietary supplement: Control drink As control, subjects are asked to consume 150 ml control drink containing equal amount of insoluble fiber (cellulose) and sugar for 28 days. In addition, on days-1 and 28, subjects will receive an acute challenge of placebo drink at our clinical facility. After 30 min. control drink intake, subjects will be given standardized breakfast corresponding to 50 g available carbohydrates.
  Interventions: Dietary Supplement: Control drink
- Berry peel drink (Experimental): Dietary supplement: Berry peel drink Subjects are asked to consume 150 ml experimental drink containing a berry peel fruit powder. In addition, on days-1 and 28, subjects will receive an acute challenge of test drink at our clinical facility. After 30 min. berry drink intake, subjects will be given standardized breakfast corresponding to 50 g available carbohydrates.
  Interventions: Dietary Supplement: Berry peel drink

INTERVENTIONS:
Dietary Supplement: Berry peel drink
  Arms: Berry peel drink
Dietary Supplement: Control drink
  Arms: Control drink

SUMMARY:
The main objective of this study is to investigate the effect of a 4-weeks intake of berry peel powder on fasting and postprandial glucose metabolism and inflammatory markers. The berry peel product will be compared with a placebo in a single-blind, cross-over design. Furthermore, inflammation-related peripheral blood mononuclear cells (PBMCs) genes expression, appetite and cognitive performance will be included as a pilot study. Investigators hypothesize that long-term consumption of polyphenols and fibres of berry peel will exhibit both direct and indirect actions in healthy overweight subjects by improvement of glucose-associated markers as well as ameliorating inflammation. Moreover, above metabolic markers will correlated with improvements in inflammation-related PBMCs genes expression, subjective appetite and cognitive performance after long-term consumption of berry peel as a source of polyphenols.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Signed informed consent
* BMI 25-30 kg/m2
* Must be able to accept plant-based foods/drinks

Exclusion Criteria:

* Below 18 years or above 40 years
* Smoking or using snuff
* vegetarian or vegan
* Stressed by venous blood sampling or previous experience of being difficult canulation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose response after acute intervention | -30, 0, 15, 30, 45, 60, 120, and 180 min after challenge meal.
  The capillary blood will be collected for glucose analysis using a glucometer.
Incremental area under curve (iAUC) blood glucose response after long-term intervention | 4 weeks
  The capillary blood will be collected for glucose analysis using a glucometer.

SECONDARY OUTCOMES:
Postprandial serum insulin response after acute intervention | -30, 0, 15, 30, 45, 60, 120, and 180 min.
  The capillary blood will be collected for insulin analysis using commercial ELISA kits
Incremental area under curve (iAUC) serum insulin response after long-term intervention | 4 weeks
  The capillary blood will be collected for insulin analysis using commercial ELISA kits
Postprandial subjective appetite rating after acute intervention | -30, 0, 15, 30, 45, 60, 120, and 180 min.
  Appetite will be assessed using standard subjective 100mm visual analogue scaled (VAS).
Incremental area under curve (iAUC) subjective appetite rating after long-term intervention | 4 weeks
  Appetite will be assessed using standard subjective 100mm visual analogue scaled (VAS).
Postprandial C-reactive protein (CRP) after acute intervention | -30, 60, 120, and 180 min.
  The venous blood will be collected for CRP analysis using ELISA commercial kits
Incremental area under curve (iAUC) of C-reactive protein (CRP) after long-term intervention | 4 weeks
  The venous blood will be collected for inflammatory analysis using ELISA commercial kits
Postprandial adiponectin after acute intervention | -30, 0, 60, 120, and 180 min.
  The venous blood will be collected for adiponectin analysis using ELISA commercial kits
Postprandial adiponectin after long-term intervention with berry peel | 4 weeks
  The venous blood will be collected for adiponectin analysis using ELISA commercial kits
Peripheral blood mononuclear cells (PBMCs) inflammatory genes expression after acute intervention | 180 min after challenge meal.
  The venous blood samples will be taken for isolation of peripheral blood mononuclear cells (PBMCs). Extracted total RNA will then be used for running quantitative-PCR.
Peripheral blood mononuclear cells (PBMCs) inflammatory genes expression after long-term intervention | -30 min. (Day-28 control); 180 min. (Day-28 control); -30 min. (Day-28 berry); 180 min. (Day-28 berry)
  The venous blood samples will be taken for isolation of peripheral blood mononuclear cells (PBMCs). Extracted total RNA will then be used for running quantitative-PCR.
Postprandial selective attention after long-term intervention | 45, 90, and 180 min after challenge meal.
  The selective attention will be assessed using a standardized software (Röd and Grön software) that measures wrong/right decisions and time of reaction when the subjects is faced with a challenging stimulus.
Postprandial interleukin-6 (IL-6) after acute intervention | -30, 60, 120, and 180 min.
  The venous blood will be collected for IL-6 analysis using ELISA commercial kits
Incremental area under curve (iAUC) of interleukin-6 (IL-6) after long-term intervention | 4 weeks
  The venous blood will be collected for IL-6 analysis using ELISA commercial kits

CONTACTS AND LOCATIONS:
Overall Officials: Angela G Batista, MSc, Study Chair — Lund University; University of Campinas; Yoghatama Cindya Zanzer, MSc, Study Chair — Lund University
Locations (1):
- Food for Health Science Centre (Medicon Village) - Lund University, Lund, Skåne County, Sweden